CLINICAL TRIAL: NCT05096949
Title: Implementing Long-Acting Cabotegravir + Rilpivirine in Arkansas Programs Utilizing Out-patient Clinics Versus In-home Visits
Brief Title: Implementing Cabenuva in Arkansas HIV Programs
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient enrollment.
Sponsor: University of Arkansas (Other)
Collaborators: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 261250
Record Dates: First submitted 2021-10-18; First posted 2021-10-27 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-01

CONDITIONS: HIV-1-infection; Medication Adherence; Satisfaction, Patient
Keywords: Delivery; Implementation; Long acting medication
MeSH Terms: conditions — Medication Adherence; Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: Cluster-randomized parallel design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Clinic visit arm (No Intervention): Patient will receive Cabenuva injection at the clinic
- Home visit arm (Experimental): Patient will receive Cabenuva injection at home
  Interventions: Other: Home visit delivery strategy

INTERVENTIONS:
Other: Home visit delivery strategy — A nurse will deliver and administer Cabenuva injection at patient's home
  Arms: Home visit arm

SUMMARY:
This study seeks to address this gap by studying two Cabenuva delivery strategies conducted at six outpatient HIV clinics in Arkansas, a Southern state with a large population of rural, poor, and African-American residents. The two delivery strategies are clinic delivery and home delivery. In the clinic delivery study arm patients will receive Cabenuva injections at the clinic (50 patients), and in the home delivery study arm patients will receive the injections at home (50 patients). The study team will follow the patients in both study arms for 10 months. After 5 months, the patients will complete a treatment satisfaction survey, and after 10 months the study team will examine clinic records to assess their medication adherence.

Secondary outcomes will include clinician perceptions of acceptability, feasibility, and appropriateness of Cabenuva delivery strategies. The study team will also collect qualitative data from patients and clinic employees to learn more in depth about their perceptions of Cabenuva, the delivery strategies, their implementation, and barriers and facilitators. Finally, the study team will estimate the costs associated with the two delivery strategies from the clinic and patient perspectives.

The data from this study provide information on what delivery strategies for long acting HIV medications offer best results, how these strategies are perceived by patients and clinicians, and how costly and feasible the strategies are to implement in practice.

DETAILED DESCRIPTION:
Good medication adherence in patients living with HIV (PLHIV) is one of the key determinants of their treatment success. Most current HIV medications are taken daily, which represents a big burden and leads to many challenges for maintaining medication adherence. These challenges are exacerbated by socio-economic factors, such as poverty, rurality, race/ethnicity, and stigma, leading to disparities in treatment and outcomes. Long acting injectable medications offer promise of reducing medication adherence burden and barriers, potentially improving the health and well-being of PLHIV, and helping limit the spread of HIV. In January 2021, FDA approved Cabenuva, the first long acting HIV medication, administered as monthly or every-2-month injections. Injectable treatment holds promise to improve treatment adherence and facilitate access to treatment for rural residents. However, it is currently not known what delivery strategies would optimize delivery of long acting HIV medications for best patient adherence and satisfaction.

This study seeks to address this gap by studying two Cabenuva delivery strategies conducted at six outpatient HIV clinics in Arkansas, a Southern state with a large population of rural, poor, and African-American residents. The two delivery strategies are clinic delivery and home delivery. In the clinic delivery study arm patients will receive Cabenuva injections at the clinic (50 patients), and in the home delivery study arm patients will receive the injection at home (50 patients). The study team will follow the patients in both study arms for 10 months. After 5 months, the patients will complete a treatment satisfaction survey, and after 10 months the study team will examine clinic records to assess their medication adherence.

Secondary outcomes will include clinician perceptions of acceptability, feasibility, and appropriateness of Cabenuva delivery strategies. The study team will also collect qualitative data from patients and clinic employees to learn more in depth about their perceptions of Cabenuva, the delivery strategies, their implementation, and barriers and facilitators. Finally, the study team will estimate the costs associated with the two delivery strategies from the clinic and patient perspectives.

The data from this study provide information on what delivery strategies for long acting HIV medications offer best results, how these strategies are perceived by patients and clinicians, and how costly and feasible the strategies are to implement in practice.

ELIGIBILITY:
Inclusion Criteria:

* Persons, 18-years old and older
* Receiving Cabenuva injections (following registered USPI) at one of the six clinics in this study
* Ability to provide informed consent
* Patients who would receive Cabenuva at home: Living within 40-miles from the three clinics randomized to the at-home arm of the study

Exclusion Criteria:

* Pregnant or breastfeeding women, or women who plan to become pregnant during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-03-07 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Medication adherence | 10 months
  Medication adherence will be quantified as a binary variable, based on whether the patient received all scheduled injections as planned or not. (As of January 2022, Cabenuva is approved for monthly and every-2-month injection schedule, and the study does not dictate which schedule the participants follow.)

SECONDARY OUTCOMES:
Patient treatment satisfaction | 5 months
  Modified version of the Satisfaction with HIV/AIDS Treatment Interview Scale (SATIS) instrument (Tran & Nguyen, 2012), with values ranging from 0 to 10 (higher scores are better).

OTHER OUTCOMES:
Clinician perceptions of acceptability | 3 months
  Modified version of Acceptability of Intervention Measure (AIM; Weiner et al., 2017), with values ranging from 1 to 5 (higher scores are better).
Clinician perceptions of appropriateness | 3 months
  Modified version of Intervention Appropriateness Measure (IAM; Weiner et al., 2017), with values ranging from 1 to 5 (higher scores are better).
Clinician perceptions of feasibility | 3 months
  Modified version of Feasibility of Intervention Measure (FIM; Weiner et al., 2017), with values ranging from 1 to 5 (higher scores are better).

CONTACTS AND LOCATIONS:
Overall Officials: Jure Baloh, PhD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: Yes
After publication, anonymized patient level data from the study may be shared with other researchers on reasonable request.

REFERENCES:
- [Background] Tran BX, Nguyen NP. Patient satisfaction with HIV/AIDS care and treatment in the decentralization of services delivery in Vietnam. PLoS One. 2012;7(10):e46680. doi: 10.1371/journal.pone.0046680. Epub 2012 Oct 5. PMID 23071611
- [Background] Weiner BJ, Lewis CC, Stanick C, Powell BJ, Dorsey CN, Clary AS, Boynton MH, Halko H. Psychometric assessment of three newly developed implementation outcome measures. Implement Sci. 2017 Aug 29;12(1):108. doi: 10.1186/s13012-017-0635-3. PMID 28851459